CLINICAL TRIAL: NCT05107349
Title: Cell Signaling, Reinnervation and Metabolism in Kennedy Disease and Amyotrophic Lateral Sclerosis (ALS)
Acronym: CERMALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D20180344; 2018-A03044-51 (Other: ANSM)
Record Dates: First submitted 2021-10-28; First posted 2021-11-04 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Amyotrophic Lateral Sclerosis; Kennedy Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Bulbo-Spinal Atrophy, X-Linked

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Other)
  Interventions: Procedure: Muscle biopsy

INTERVENTIONS:
Procedure: Muscle biopsy — A motor point biopsy of deltoid muscle will be carried out at the time of inclusion using a standardized procedure, as routinely performed. Muscle samples will be removed from the deltoid muscle by open biopsy under local anaesthesia. The region containing NMJs will be determined by the small twitch provoked by the tip of the scalpel on the surface of the muscle fascicles.

SUMMARY:
Amyotrophic lateral sclerosis (ALS), is a rapidly progressive neurodegenerative disorder, usually leading to death from respiratory failure in 3-5 years. Riluzole, the only drug currently available, only modestly prolongs survival and does not improve muscle strength or function. In ALS, loss of functional motor neurons is initially compensated for by collateral reinnervation and strength is preserved. In the majority of ALS patients, as the disease progresses, compensation fails leading to progressive muscle weakness. Conversely, in long-term ALS survivors, slow functional decline is correlated with their ability to maintain a successful compensatory response to denervation over time. Compensatory collateral reinnervation is thus essential for functional motor preservation and survival, and elucidation of the molecular mechanisms involved is crucial to help identify new therapeutic targets. Energy metabolism and glucose homeostasis modifications also influence disease clinical course but the mechanisms by which they contribute to the progression of ALS are unknown. Weight loss is an independent negative prognostic factor for survival and, by contrast, ALS risk and progression are decreased in individuals with high body mass index and non-insulin-dependent diabetes mellitus. Insulin shares many common steps in its signaling pathways with insulin-like growth factor 1 (IGF-1), and is thus at the interface between glucose homeostasis regulation and maintenance of muscle mass. However, the contribution of insulin signaling to preservation of muscle innervation and function in ALS has never been investigated.

With this study, we aim to determine the role of insulin signaling pathways in maintenance of collateral reinnervation and muscle function in ALS. We will also investigate the link with the disease-modifying effect of metabolic and glucose homeostasis perturbations, by identifying the contribution of metabolic profiles to preservation of skeletal muscle innervation and motor function in patients with ALS. For this purpose, we will determine the whole-body and skeletal muscle metabolic profiles of 20 patients with ALS and correlate these results to collateral reinnervation ability quantified on muscle biopsy specimens. For each patient, we will use both clinical and electrophysiological methods to evaluate motor function and motor neuron loss over time. Body composition, insulin secretion, insulin resistance level and serum concentrations of IGF-1 axis components will be determined. A motor point muscle biopsy will be performed for morphological analysis of neuromuscular junctions and quantification of innervation by confocal microscopy. Activation of insulin/IGF-1 canonical signaling pathways and metabolic pathways of glucose homeostasis will be quantified in muscle specimens. Skeletal muscle and whole-body metabolic parameters will be analyzed together and correlated with clinical assessment of motor function, electrophysiological data, and innervation quantification results. For comparison, 10 healthy subjects of similar age and 10 patients with spinal and bulbar muscular atrophy - a slowly progressive motor neuron disorder with maintenance of effective collateral reinnervation - will be used as controls. This study will be the first to address the question of the contribution of insulin signaling pathways and metabolic profiles in maintenance of muscle reinnervation and function in ALS patients. The molecular mechanisms identified will be new targets for future treatments promoting compensatory reinnervation and slowing disease progression in ALS. Ultimately, this translational project could have a significant therapeutic impact in disorders with muscle denervation and collateral reinnervation as a compensatory mechanism, such as spinal muscle atrophy or peripheral neuropathies.

DETAILED DESCRIPTION:
In amyotrophic lateral sclerosis (ALS), loss of functional motor neurons is initially compensated for by collateral reinnervation but, as the disease progresses, compensation usually fails leading to progressive muscle weakness. Conversely, in long-term ALS survivors, slow functional decline is correlated with their ability to maintain a successful compensatory response to denervation over time. The molecular mechanisms by which compensatory reinnervation, a crucial process for function and survival, is maintained over time remains to be elucidated. We have previously shown that muscle factors may be involved in maintenance of muscle innervation and function in ALS long-term survivors (Bruneteau et al.,2013). Energy metabolism and glucose homeostasis modifications also influence disease clinical course but the mechanisms by which they contribute to ALS progression are unknown. Insulin signaling cascades share many common steps with Insulin-like Growth Factor-1 (IGF-1) signaling pathways, and link maintenance of muscle mass with glucose and energy metabolism which are both connected to ALS progression. Our working hypothesis is that insulin signaling pathways play a major role in maintaining collateral reinnervation and muscle function in ALS. To comfort this hypothesis, we will quantify innervation in muscle specimens obtained from ALS patients and correlate these results to the level of activation of insulin main signaling pathways and expression of key determinants of glucose metabolism. These data will be analyzed together with evaluation of motor function and motor neuron loss over time, to understand how insulin signaling and glucose homeostasis influence disease progression. To decipher how energy and glucose metabolism are involved in preservation of a high level of collateral reinnervation over time, results obtained in ALS patients will be compared to those of normal subjects of similar age and patients with spinal and bulbar muscular atrophy (SBMA).

PATIENTS EVALUATION

1. Clinical evaluation

   * Characteristics of patients
   * Patient characteristics will be reviewed at the time of inclusion: personal or familial history of medical conditions, age at onset, localization of onset (limb or bulbar), concomitant medications including riluzole.
   * Disease evaluation will be performed at baseline, 3 months, 6 months and 12 months:
   * Functional impairment will be assessed using the revised ALS Functional Rating Scale (ALSFRS-R), a 12-item scale that rates the performance of activities of daily living. Signs and symptoms range from 4 (normal function) to 0 (unable to attempt the task) (Cedarbaum et al.,1999). Twelve functions are listed, including: speech, salivation and swallowing for bulbar involvement; writing, feeding, dressing, turning in bed, walking and climbing stairs for upper and lower limbs involvement; respiratory function.
   * Muscle strength will be measured on 28 muscles by manual muscle testing according to the grading system of the Medical Research Council.
2. Laboratory tests

   * The routine biological tests, including platelet count and coagulation test will be performed at baseline
   * For all patients, genetic screening of all major ALS-associated genes will be performed at the time of inclusion (including C9ORF72, SOD1, TARDBP, FUS, UBQLN2, TBK1 genes to date and any novel major ALS-linked gene that could be discovered).
   * Respiratory function will be assessed at baseline, M6 and M12 as part of the routine follow-up procedure in the ALS center, including vital capacity expressed as a percentage of the predicted normal vital capacity, arterial blood gas analysis for determination of partial pressure of arterial oxygen and carbon dioxide, and nocturnal pulse oximetry (oxyhemoglobin saturation).
3. Surface EMG procedure and motor unit number index (MUNIX) measurement Surface EMG evaluation of neuromuscular function will be performed in all patients at baseline. The standardized EMG protocol will include motor nerve conduction studies of upper and lower limbs, and repetitive nerve stimulation studies for assessment of neuromuscular transmission on the spinal accessory nerve, the axillary nerve, the ulnar nerve and the radial nerve of both upper limbs. MUNIX measurement will be performed on deltoid and biceps brachii muscles, at baseline, 3 months, 6 months and 12 months.
4. Assessment of nutritional status and general metabolic profile

Assessment of nutritional status and general metabolic profile will be performed at baseline for the two groups of patients and will include:

* Data collection for weight, height, BMI determination, waist and hip circumference (waist/hip ratio calculation), nutrient intake
* Measurements of body composition with whole body Dual X-Ray Absorptiometry (DEXA)
* Assessment of resting energy expenditure (indirect calorimetry)
* Evaluation of insulin secretion and insulin resistance with measurement of glucose and insulin levels before and 30 mn after ingestion of a standardized liquid meal test. Insulin resistance and insulin secretion will be evaluated by calculation of HOMA-IR (insulin resistance index) and insulin secretion will be evaluated by calculation of HOMA-B (insulin secretion index) and insulinogenic index.
* Determination of serum concentrations of IGF-1 axis components.

MOTOR-POINT MUSCLE BIOPSY PROCEDURE For all patients, muscle samples will be removed from the deltoid muscle by open biopsy under local anaesthesia for all patients. The region containing NMJs will be determined by the small twitch provoked by the tip of the scalpel on the surface of the muscle fascicles. For healthy control subjects, biopsy specimens of deltoid muscle will be obtained during shoulder surgery for joint or bone disease.

The presence of NMJs on a longitudinal strip of the biopsy specimen will be confirmed using the classic Koelle method revealing cholinesterase activity (Koelle and Friedenwald ,1949). Each biopsy specimen will be sub-divided into several muscle fragments. For confocal imaging study of the morphology of NMJs, muscle samples will be fixed in 4% paraformaldehyde. For electron microscopy study of NMJ ultrastructure, thin strips of muscle from the sample will be fixed in a mixture of paraformaldehyde 2% and glutaraldehyde 2.5%. Several muscle fragments will be fresh frozen in isopentane for histological, biochemical, and molecular studies.

ELIGIBILITY:
Inclusion Criteria:

* Twenty patients with ALS, including 10 patients with more than 5 years of disease progression without requiring respiratory support or gastrostomy feeding. All ALS patients will fulfill the following inclusion criteria:
* Aged 18 to 80 (inclusive)
* Possible, probable (clinically or laboratory) or definite ALS according to the revised version of the El Escorial World Federation of Neurology criteria (Brooks et al.,2000)
* Ten patients with Spinal-bulbar muscular atrophy (SBMA), aged 18 to 80
* Ten healthy subjects: Control muscle specimens (deltoid) will be obtained from 10 adult patients (aged 18-80) without neuromuscular disease, undergoing shoulder surgery for local joint or bone disease in the local department of orthopaedic surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Quantification of neuromuscular junctions innervation | At 15 days after inclusion visit
  Quantification of innervation by confocal microscopy will be performed by classifying neuromuscular junctions observed in each biopsy specimen according to the relationship between the intrasynaptic axonal branches and the postsynaptic membrane in four categories: "normal", "denervated", "partially innervated", or "reinnervated"

SECONDARY OUTCOMES:
Level of the main components of the insulin/IGF-1 system | 12 months
Correlations between metabolic profiles and muscle function | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gaelle Bruneteau, MD, PhD, Principal Investigator — APHP - Hôpital Pitié-Salpêtrière
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.